CLINICAL TRIAL: NCT04537377
Title: A Phase I/II, Multicenter, Non-randomized, Open Label, Adaptive Design, 5-year Follow-up, Single Dose-escalation Study of VTX-801 in Adult Patients With Wilson's Disease
Brief Title: A Phase I/II Study of VTX-801 in Adult Patients With Wilson's Disease
Acronym: GATEWAY
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vivet Therapeutics SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VTX-801_CLN_001; 2020-000963-22 (EudraCT Number)
Record Dates: First submitted 2020-08-19; First posted 2020-09-03 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VTX-801 (Experimental)
  Interventions: Genetic: VTX-801

INTERVENTIONS:
Genetic: VTX-801 — The investigational medicinal product (VTX-801) is a replication-deficient recombinant adeno-associated viral vector (rAAV) consisting of an AAV liver tropic capsid containing a single-stranded DNA genome carrying a shortened version of the ATP7B gene (ATP7B-minigene).
  After reconstitution VTX-801 will be administered as a single dose intravenous (IV) administration per patient, at up to 3 different dose levels.

SUMMARY:
The objectives of this clinical trial are to assess, for up to 5 years, the safety, tolerability and pharmacological activity of a single ascending doses of VTX-801, a gene therapy, administered intravenously (IV) to adult patients with Wilson's Disease prior to and following background WD therapy withdrawal.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female aged 18 and 65 years inclusive
* Confirmed diagnosis of WD
* Treated for WD according to international recommendations with no current evidence for inadequate treatment
* Stable WD for ≥ 1 year, defined as: (i) No significant change in neurologic examination and in status of mood disorder and (ii) Stable laboratory parameters used to assess copper metabolism

Main Exclusion Criteria:

* ALT level ≥ 2 ULN that is not readily explained by extrinsic factors
* Total bilirubin > 1.5 x ULN in the absence of proven Gilbert's syndrome; in case of Gilbert's syndrome, direct bilirubin > ULN
* INR > 1.2
* Any signs of liver cirrhosis decompensation, including gastrointestinal bleed within 6 months (24 weeks) prior to screening/enrollment visit
* Patient has moderate or severe renal impairment defined as eGFR CKD-EPI < 60 mL/min/1.73 m2, or patient has nephritis or nephrotic syndrome
* Any history or current evidence of HIV-1, HIV-2, HTLV 1, or HTLV-2 infection
* Any history or current evidence of hepatitis B infection
* Any history of hepatitis C infection, unless previous viral RNA assays in two samples, collected at least 6 months apart, are negative
* Positive QuantiFERON®-TB Gold tuberculosis test result
* Any concomitant disorder/condition - including hepatic disorders - or treatment possibly interfering with the conduct or evaluation of the study
* Any history of diabetes
* Pregnancy or breastfeeding
* Body Mass Index ≥ 35 kg/m2

Other protocol defined Inclusion/ Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2029-06-18 (Estimated)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - UC Davis Medical Center, Sacramento, California
  - Yale University School of Medecine, New Haven, Connecticut
  - Advent Health, Orlando, Florida
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Aarhus University Hospital, Aarhus, Denmark
- Germany (2):
  - University Hospital Essen, Essen
  - Universitätsklinikum Tübingen (UKT), Tübingen
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was prematurely terminated by the Sponsor for futility reasons, after insufficient pharmacodynamic response in cohorts 1 and 2. No further patient enrollment occurred after this date. The 4 treated patients entered the long-term follow-up (LTFU) up to 5 years post injection, thus 2 sites remain active.
  An abbreviated CSR was issued including all data until early termination (an average of 1 year). The LTFU results will be provided in a separate addendum at the end of 2029.
Groups:
- VTX-801 5E12 VG/kg: Cohort 1: Patients received a single IV infusion of VTX-801 at 5E12 VG/kg and with a 5-year follow-up.
- VTX-801 1.5E13 VG/kg: Cohort 2: Patients received a single IV infusion of VTX-801 at 1.5E13 VG/kg and with a 5-year follow-up.
Period: Overall Study
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg
Started | 2 | 2
End of Primary Completion Period | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Long term follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (17.68) | 32.0 (18.38) | 34.3 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Smoking History [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 2 | 2 | 4
Alcohol Consumption [Count of Participants; unit: Participants]
  Yes current | 1 | 0 | 1
  Yes former | 1 | 0 | 1
  No | 0 | 2 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (2.0) | 29.7 (4.64) | 27.6 (3.83)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Profile (Including Treatment-emergent Adverse Events (TEAE)) - Number of Participants
Description: AEs will be summarized based on the date of onset for the event. Number of treatment-emergent AEs will be provided by SOC and PT, by dose cohort and overall.
Time Frame: through primary completion visit, an average of 1 year
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg
Number analyzed (Participants) | 2 | 2
participants
  Treatment-emergent AEs | 2 | 2
  Deaths | 0 | 0
  SAEs | 0 | 1
  AEs leading to discontinuation | 0 | 0
  TEAE meeting any stopping rule | 2 | 2

2. Secondary Outcome: Free Serum Cu
Description: Free serum Cu will be summarized descriptively for all patients by dose cohort and planned visit, for absolute values and changes from baseline.
Time Frame: through primary completion visit, an average of 1 year
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg
Number analyzed (Participants) | 2 | 2
umol/L
  Absolut value | 1.080 (0.6930) | 0.620 (0.1556)
  CFB | 0.115 (0.3465) | -0.225 (0.3182)

3. Secondary Outcome: Total Serum Cu
Description: Total serum Cu will be summarized descriptively for all patients by dose cohort and planned visit, for absolute values and changes from baseline.
Time Frame: through primary completion visit, an average of 1 year
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg
Number analyzed (Participants) | 2 | 2
umol/L
  Absolut value | 2.595 (0.3889) | 5.185 (5.4094)
  CFB | 0.700 (0.5091) | 1.185 (1.4354)

4. Secondary Outcome: 24-hour Urinary Cu
Description: 24-hour urinary Cu will be summarized descriptively for all patients by dose cohort and planned visit, for absolute values and changes from baseline.
Time Frame: through primary completion visit, an average of 1 year
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: mcg/24hr
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg
Number analyzed (Participants) | 2 | 2
mcg/24hr
  Absolut value | 78.0 (5.66) | 85.5 (61.52)
  CFB | -7.0 (1.41) | 7.0 (22.63)

5. Secondary Outcome: Serum Ceruloplasmin Activity (Enzymatic Assay)
Description: Serum ceruloplasmin will be summarized descriptively for all patients by dose cohort and planned visit, for absolute values and changes from baseline.
Time Frame: through primary completion visit, an average of 1 year
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: nmol Fe2+/min/mL
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg
Number analyzed (Participants) | 2 | 2
nmol Fe2+/min/mL
  Absolut value | 10.75 (0.495) | 42.80 (46.810)
  CFB | 1.05 (1.344) | -27.40 (39.174)

6. Secondary Outcome: VTX-801 Responder Status
Description: The number of Responders and Insufficient-Responders will be summarized by dose cohort and planned visit, with response to treatment. Responder status was assessed using radiocopper blood PK results and other cold copper parameters if needed.
Time Frame: At Week 12 and Week 36
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg
Number analyzed (Participants) | 2 | 2
Participants
  W12: Responder | 0 | 0
  W12: Insufficient Responder | 2 | 2
  W12: Not assessed | 0 | 0
  W36: Responder | 0 | 0
  W36: Insufficient Responder | 2 | 0
  W36: Not assessed | 0 | 2

ADVERSE EVENTS:
Time Frame: From Baseline through primary completion visit (an average of 1 year)
Arm/Group | VTX-801 5E12 VG/kg | VTX-801 1.5E13 VG/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VTX-801 5E12 VG/kg (N=2) | VTX-801 1.5E13 VG/kg (N=2)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VTX-801 5E12 VG/kg (N=2) | VTX-801 1.5E13 VG/kg (N=2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 1 (2) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 2 (7) | 2 (2)
Lymphocyte Count Decreased (Investigations) | 1 (2) | 1 (2)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (3)
Body Temperature Increased (Investigations) | 0 (0) | 1 (1)
Drug Level Increased (Investigations) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0)
Urine Copper Increased (Investigations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Brain Fog (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Kayser-Fleischer Ring (Eye disorders) | 1 (1) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to futility and not for safety reasons, because the VTX-801 pharmacodynamics effects observed in the first 4 patients at the first 2 dose levels tested were insufficient to allow withdrawal of the SoC.

Due to the early study termination and limited data, no conclusions can be drawn regarding the predefined objectives. The safety results were consistent with the expected safety profile for VTX-801. No new safety issues were observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor can request deletions to Confidential Information to the extent such deletion does not preclude the complete and accurate presentation and interpretation of the Study results.

DOCUMENTS (2):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT04537377/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT04537377/SAP_001.pdf